CLINICAL TRIAL: NCT05374382
Title: The Effects of a Lower Limb Strengthening Training Program During Prehabilitation Prior to ACL Surgery on Lower Limb Structure and Function : a Randomized Clinical Trial
Brief Title: A Prehab Strengthening Program Prior to ACL Surgery on Lower Limb Structure and Function
Acronym: ACL-Strong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Nantes (Other)
Responsible Party: Principal Investigator, Guillaume Le Sant, Guillaume Le Sant, PhD,PT. Physiotherapist and Researcher, Université de Nantes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACL-Strong
Record Dates: First submitted 2022-05-02; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: ACL Injury
Keywords: rehabilitation; strengthening; physiotherapy; atrophy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Atrophy | interventions — Resistance Training; Congresses as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strengthening (Experimental): Participants received a 9-weeks strengthening-based prehabilitation program before ACL reconstruction, followed by a standardized post-operative rehabilitation program
  Interventions: Behavioral: Strengthening
- Conventional (Active Comparator): Participants received a 9-weeks conventional prehabilitation program (targeting pain knee mobility) before ACL reconstruction, followed by a standardized post-operative rehabilitation program
  Interventions: Behavioral: Conventional
- Control (No Intervention): No prehabilitation program Participants received only a standardized post-operative rehabilitation program

INTERVENTIONS:
Behavioral: Strengthening — 3x/w, 9 wks supervised strengthening program, during prehabilitation to ACL surgery
  Arms: Strengthening
Behavioral: Conventional — Participants received a 9-weeks conventional prehabilitation program (targeting pain knee mobility) before ACL reconstruction, followed by a standardized post-operative rehabilitation program
  Arms: Conventional

SUMMARY:
Atrophy and weakness are ubiquitous after a ACL rupture and associated with a worsened long-term recovery of individual capacities, despite surgery and rehabilitation. Preoperative rehabilitation (prehab) is believed to prepare patients for surgery and post-operative rehabilitation. However, prehab programs are highly variable, and do not always aim to develop/maintain neuromuscular parameters.

The purpose of this study is to assess the effects of a lower limb strengthening training program during prehab prior to ACL Surgery on lower limb structure and function.

DETAILED DESCRIPTION:
Recruited participants will be randomly allocated to one of the three groups of participants constituted in this study.

The two first groups will receive prehabilitation prior to ACL reconstruction (differing in program type). All participants will receive standardized post-surgery rehabilitation (based on international recommandations).

ELIGIBILITY:
Inclusion Criteria:

* age : 18 to 55
* first episode of ACL injury
* having a planed ACL reconstruction
* volunteer to participate

Exclusion Criteria:

* age : <18 or >55
* previous episode of ACL injury/reconstruction
* no ACL reconstruction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle strength of the knee muscles | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Maximal muscle strength of knee flexors/extensors will be assessed using isokinetic dynamometer, and extension and flexion torques during a maximum voluntary contraction (MVC).
  Unit : Newton meter (Nm)
Change in muscle volume of the knee muscles | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Muscle volume of the knee muscles (hamstring and quadriceps) will be assessed using 3D ultrasound imaging, at rest in a prone (hamstring) or supined (quadriceps) position.
  Unit : millimeters (mL)
Change in the stiffness of knee muscles | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  An index of muscle stiffness will be assessed via the shear modulus using ultrasound shear wave elastography, at rest in a prone (hamstring) or supined (quadriceps) position.
  Unit : kiloPascals (kPa)
Change in lower limb function | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Single leg hop test. Participants will be instructed to jump as far as possible on a single leg, without losing balance and landing firmly. The distance is measured from the start line to the heel of the landing leg.
  Unit : centimeters (cm)
Change in patient's opinion about the knee and associated problems | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Patient's self-related opinion about symptoms and activity will be assessed using the International Knee Documentation Committee Subjective Knee Form (IKDC).The IKDC is consisted of 10 questions.
  Unit : score, scaled between 0 (=bad) and 100 (= good function)
Change in patient's opinion to return to sport | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Patient's self-related opinion out the impact of returning to sport will be assessed using the Anterior Cruciate Ligament - Return to Sport after Injury (ACL-RSI) questionnaire.
  The ACL-RSI consists of 12 questions. Unit : score, scaled between 0 (=bad) and 100 (= more psychologically ready to return to sport)

SECONDARY OUTCOMES:
Health consumption | week 0 (baseline); week 9 (post-intervention, short term) ; 6 months after the surgery (post-intervention, mid-term) and 12 months after the surgery (post-intervention, long-term)
  Drugs intakes, dates of physiotherapy/medical consultations, date of return to work will be assessed through a diary
  Unit : self-reported date, in a paper diary

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Le Sant, PhD, PT, Principal Investigator — Université de Nantes
Locations (1):
- Université de Nantes - MIP UR 4334 (Motricity, Movement, Interactions), Nantes, France

IPD SHARING:
Plan to Share IPD: No